CLINICAL TRIAL: NCT05663996
Title: The Effect of St. John's Wort Oil on Pain Intensity and Physical Functions in People With Knee Osteoarthritis: a Qualitative and Randomized Placebo-controlled Trial
Brief Title: St. John's Wort Oil on Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Deniz Zeynep SÖNMEZ, assistant professor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TDK-2017-7629
Record Dates: First submitted 2022-12-02; First posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Osteoarthritis, Knee; Pain
Keywords: osteoarthritis; pain; St. John's Wort oil; physical function; nursing
MeSH Terms: conditions — Osteoarthritis, Knee; Pain; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: The study was conducted using a pre-test and post-test, randomized controlled trial pattern and semi-structured in-depth interview method of qualitative research.
Who Masked: Participant
Masking Description: Patients diagnosed with osteoarthritis by a physical therapy and rehabilitation specialist according to ACR criteria were randomized into the study by the University Biostatistics Unit.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- St. John's Wort oil (Experimental): Experimental group participants were treated with St. John's Wort oil.
  Interventions: Other: locally applied to the skin
- Olive Oil (Placebo Comparator): Control group participants were treated with olive oil.
  Interventions: Other: locally applied to the skin

INTERVENTIONS:
Other: locally applied to the skin — Applying St John's wort oil locally on the knee three times a day for three weeks.
  Arms: St. John's Wort oil
Other: locally applied to the skin — Applying olive oil locally on the knee three times a day for three weeks.
  Arms: Olive Oil

SUMMARY:
This study investigated the effect of St. John's Wort oil on pain intensity and physical functions in people with knee osteoarthritis. This study adopted a randomized, placebo-controlled, and qualitative mixed design. The sample consisted of 60 patients randomized into intervention (n=30) and placebo control (n=30) groups. The experimental group participants were treated with St. John's Wort oil three times a week for three weeks, while the placebo control group participants were treated with olive oil three times a week for three weeks. Quantitative data were collected using a patient identification form, the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), and the Visual Analogue Scale (VAS). Qualitative data were collected through semi-structured interviews. .

DETAILED DESCRIPTION:
This study adopted a randomized, placebo-controlled, and qualitative mixed design. Qualitative data were collected using a semi-structured interview questionnaire.

The study was conducted in the physical therapy and rehabilitation outpatient clinic of a public hospital in Türkiye. The study population consisted of all patients admitted to the outpatient clinic for osteoarthritis-related pain. The data collection process continued from December 2017 to August 2018 and was reported in accordance with the Consolidated Standards of Reporting Trials (CONSORT) guidelines. A pilot study was conducted with five patients before data collection.

Patients diagnosed with osteoarthritis by a physical therapy and rehabilitation specialist according to ACR criteria were randomized into the study by the University Biostatistics Unit. The initial sample consisted of 72 patients divided into intervention (n=36; St. John's wort oil) and placebo control (n=36; olive oil) groups. However, six experimental group participants were excluded because they either could not be contacted on the phone during the follow-ups (n=4) or stated that they would be out of town for a long time (n=2). Six control group participants were also excluded because they either could not be contacted on the phone during the follow-ups (n=3), did not want to keep up with the intervention (n=1), or wanted to withdraw from the study (n=2). Therefore, the final sample consisted of 30 experimental and 30 control group participants.

ELIGIBILITY:
Inclusion Criteria:

* being literate,
* planning no pregnancy during the study,
* not being pregnant,
* having been diagnosed with knee osteoarthritis according to ACR (American College of Rheumatology),
* having had knee pain for the past month,
* needing analgesics for more than 15 days in a month,
* having osteoarthritis-related knee pain despite routine treatment with analgesics,
* having a VAS score of ≥ 4 on one knee,
* speaking Turkish,
* having no communication problems, and
* volunteering

Exclusion Criteria:

* Pregnant,
* Having a physical disability in the area where the application will be made,
* Having any skin disease in the area to be treated,
* Having large scar tissue in the area to be treated,
* Having a history of physical trauma in the last three months in the area to be treated,
* Having any peripheral vascular disease in the area to be treated,
* Having inflammatory joint disease,
* Having a history of rheumatoid arthritis and fibromyalgia,
* Using any complementary and integrative (integrated) health application in the last three months,
* Those who have undergone intra-articular treatment in the last three months,
* Receiving pain blocking treatment in the last year,
* Receiving physical therapy in the last three months and during the application,
* Patients with 2 or more pain in the other knee according to the VAS scale were not included in the study.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-12-25 (Actual); Primary Completion 2018-08-06 (Actual); Study Completion 2018-08-06 (Actual)

PRIMARY OUTCOMES:
WOMAC Scale | Change from baseline score at the end of the third week
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a health status scale assessing osteoarthritis-related disability. WOMAC was developed (1982) and revised (1998) by Bellamy et al. The index consists of 24 items rated on a five-point Likert-type scale. The index has three subscales: pain (five items), stiffness (two items), and physical function (17 items). WOMAC can detect significant health status changes following various pharmacological, surgical, and physical therapy interventions. The instrument has been adapted into many languages. The total score of the "pain" subscale ranges from 0 to 20. The total score of the "stiffness" subscale ranges from 0 to 8. The total score of the "physical function" subscale ranges from 0 to 68. Higher scores indicate more symptoms and physical limitations.
Visual Analog Scale | change in baseline scores at the end of the third week.
  The Visual Analog Scale was developed by Price et al. (1983). It is an easy-to-use and reliable scale used to convert some values that cannot be measured numerically into numbers. The VAS is a 10 cm long horizontal or vertical line with anchor statements "no pain or pain at its least" at the left-most end and "unbearable pain or worst pain imaginable" at the right-most end. The participant marks a point on the line that best represents their pain level. The distance of the mark to the left end is measured with a ruler. This distance, usually measured in millimeters, is reported and recorded as "points.

CONTACTS AND LOCATIONS:
Locations (1):
- Osmaniye Korkut Ata University, Osmaniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barthel HR, Haselwood D, Longley S 3rd, Gold MS, Altman RD. Randomized controlled trial of diclofenac sodium gel in knee osteoarthritis. Semin Arthritis Rheum. 2009 Dec;39(3):203-12. doi: 10.1016/j.semarthrit.2009.09.002. PMID 19932833
- [Background] Kooshki A, Forouzan R, Rakhshani MH, Mohammadi M. Effect of Topical Application of Nigella Sativa Oil and Oral Acetaminophen on Pain in Elderly with Knee Osteoarthritis: A Crossover Clinical Trial. Electron Physician. 2016 Nov 25;8(11):3193-3197. doi: 10.19082/3193. eCollection 2016 Nov. PMID 28344755
- [Background] Altındağ, Ö., Sırmatel, Ö., & Tabur,H. (2006). Demographic features and relation with clinical parameters in patients with knee osteoarthritis. Harran Üniversitesi Tıp Fakültesi Dergisi, 3(2), 62-66
- [Background] Tütün, Ş., Altın, F., Özgönenel, L, & Çetin, E. (2010). Demographic characteristics in patients with knee osteoarthritis and relationship with obesity, Age, Pain and Gender. İstanbul Med J, 11(3), 109-112.
- [Background] Gümüş, K. & Ünsal A. (2014). Evaluation of daily living activities of the individuals with osteoarthritis. Turkish Journal of Osteoporosis, 20,117-24. http://doi:10.4274/tod.93723
- [Background] Bellamy N, Buchanan WW, Goldsmith CH, Campbell J, Stitt LW. Validation study of WOMAC: a health status instrument for measuring clinically important patient relevant outcomes to antirheumatic drug therapy in patients with osteoarthritis of the hip or knee. J Rheumatol. 1988 Dec;15(12):1833-40. PMID 3068365
- [Background] İnan, Ç., & Kıyak, E., (2014) The effect of hot and cold application on pain, stiffness and physical function in patients with knee osteoarthritis. Hemşirelikte Araştırma ve Geliştirme Dergisi, 16(2), 1-10.
- [Background] Chen L, Li D, Zhong J, Qiu B, Wu X. Therapeutic Effectiveness and Safety of Mesotherapy in Patients with Osteoarthritis of the Knee. Evid Based Complement Alternat Med. 2018 Jan 4;2018:6513049. doi: 10.1155/2018/6513049. eCollection 2018. PMID 29507592
- [Background] Cheung C, Wyman JF, Bronas U, McCarthy T, Rudser K, Mathiason MA. Managing knee osteoarthritis with yoga or aerobic/strengthening exercise programs in older adults: a pilot randomized controlled trial. Rheumatol Int. 2017 Mar;37(3):389-398. doi: 10.1007/s00296-016-3620-2. Epub 2016 Dec 2. PMID 27913870
- [Background] Tuzun EH, Eker L, Aytar A, Daskapan A, Bayramoglu M. Acceptability, reliability, validity and responsiveness of the Turkish version of WOMAC osteoarthritis index. Osteoarthritis Cartilage. 2005 Jan;13(1):28-33. doi: 10.1016/j.joca.2004.10.010. PMID 15639634
- [Background] Price DD, McGrath PA, Rafii A, Buckingham B. The validation of visual analogue scales as ratio scale measures for chronic and experimental pain. Pain. 1983 Sep;17(1):45-56. doi: 10.1016/0304-3959(83)90126-4. PMID 6226917
- [Background] Kelly AM. Does the clinically significant difference in visual analog scale pain scores vary with gender, age, or cause of pain? Acad Emerg Med. 1998 Nov;5(11):1086-90. doi: 10.1111/j.1553-2712.1998.tb02667.x. PMID 9835471
- [Background] Williamson A, Hoggart B. Pain: a review of three commonly used pain rating scales. J Clin Nurs. 2005 Aug;14(7):798-804. doi: 10.1111/j.1365-2702.2005.01121.x. PMID 16000093
- [Background] Sentürk, S., Tasci, S. (2021). The effects of ginger kidney compress on severity of pain and physical functions of individuals with knee osteoarthritis: A Randomized Controlled Trial International Journal of Traditional and Complementary Medicine Research, 2(2): 83-94. http://doi:10.53811/ijtcmr.972187
- [Background] Dogan N, Goris S, Demir H. [Levels of pain and self-efficacy of individuals with osteoarthritis]. Agri. 2016 Jan;28(1):25-31. doi: 10.5505/agri.2015.30085. Turkish. PMID 27225609